CLINICAL TRIAL: NCT04009473
Title: Platelet Rich Plasma Ovarian in Vitro Activation and Stem Cells Transplantation In Women With Ovarian Failure
Brief Title: Stem Cell Therapy and Growth Factor Ovarian in Vitro Activation
Acronym: SEGOVA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Forever Young d.o.o. (Other)
Collaborators: Medigroup Health System, Jevremova hospital (Other); Saint James Hospital Malta (Unknown); Re-medika Hospital Skoplje (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB No 63/295/2015
Record Dates: First submitted 2019-06-29; First posted 2019-07-05 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Menopause; Menopause Ovarian Failure; Ovarian Failure; Premature Ovarian Failure; Premature Ovarian Failure 1; Premature Ovarian Failure 2A; Premature Ovarian Failure 2B; Premature Ovarian Failure 3; Premature Ovarian Failure 4; Premature Ovarian Failure 5; Premature Ovarian Failure 6; Premature Ovarian Failure 7; Premature Ovarian Failure 8; Premature Ovarian Failure 9; Premature Ovarian Failure 10; Premature Ovarian Failure 11; Premature Ovarian Failure 12; Premature Ovarian Failure 13; Premature Ovarian Failure 14; Ovarian Insufficiency; Ovarian Failure Secondary; Ovarian Failure, Premature; Ovarian Insufficiency, Primary; Menopause, Premature
Keywords: platelet rich plasma; growth factors; stem cells; bone marrow; in vitro activation; ovarian cortex transplantation; hippo signalling pathway
MeSH Terms: conditions — Primary Ovarian Insufficiency; Premature Ovarian Failure 2a; Premature Ovarian Failure 2b; Premature Ovarian Failure 3; Ovarian Dysgenesis 2; Premature Ovarian Failure 5; Premature Ovarian Failure 6; Premature Ovarian Failure 7; Menopause, Premature

STUDY DESIGN:
Intervention Model Description: Pre-post study design:
  A study group receives the intervention, and the changes in parameters were measured and compared before and after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- SEGOVA Intervention Group (Experimental): Intervention group of 50-100 patients with ovarian failure would be subjected to a three-day procedure named SEGOVA: bone marrow derived StEm cell treatment, Growth factor incubation and Ovarian In Vitro Activation. After the procedure, one year follow up of hormones measurements (follicle stimulating hormone (FSH), luteinizing hormone (LH),estradiol (E2), progesterone (PG) and anti-mullerian hormone (AMH)) and follicle counts would be established. In patients with oocytes retrieved after SEGOVA procedure, standard In Vitro Fertilization protocol would be performed. The fertilization, cleavage and clinical pregnancy rate will be monitored.
  Interventions: Combination Product: SEGOVA procedure

INTERVENTIONS:
Combination Product: SEGOVA procedure — SEGOVA procedure includes - Stem cell therapy, G - Growth factor Platelet Plasma Rich therapy and in Vitro Activation of the ovaries.

SUMMARY:
SEGOVA procedure includes - Stem cell therapy, G - Growth factor Platelet Plasma Rich therapy and in Vitro Activation of the ovaries.

DETAILED DESCRIPTION:
The current study seeks to demonstrate how integrative ovarian rejuvenation program called SEGOVA influence the restoration of hormone stability and increase in the number of follicles in ovarian failure patients. The recruitment of patients and data collection would be performed at three sites: The Special Hospital Jevremova Belgrade, Saint James Hospital Malta, and Remedica Skopje Hospital, Macedonia. A 50-100 of Infertile women with ovarian failure will be included in the period between July 2019 - December 2021. The patients would be coded when entering the program, and all personal information would be protected. Information about medical treatment and background will be held on both paper and electronic case report forms.The result of the procedure will be maintained in the research database with blinding to clinical physician that will perform post procedure follow-up of those patients. In case of a complication, possibly related to treatment, the case will be unblinded.

The first day of procedure, autologous platelet rich plasma (PRP) is obtained from 100-120 mL of whole blood. After separation 4 mL of PRP is obtained. Concentration of platelets is optimised on 6-8x baseline and 2-3x leucocytes baseline. For activation of PRP autologous thrombin is used in ratio 1:10.

On the same day the laparoscopic cortical resection of the ovary is performed in standard technique. Ovarian cortex sample is minced in a petri dish.The volume of activated PRP (4 mL) is mixed with ovarian fragments and incubated for the next 48h at 37℃ and 5% CO2. After 48h, the bone marrow sampling from tibia under general anesthesia is performed to obtain bone marrow. After centrifugation the Bone Marrow Aspirate Concentrate (BMAC) with nucleated cells is obtained (3 +/- 1,5 mL).

Finally, after the 48h has passed from ovarian cortex tissue incubation, fragmented tissue of the ovary with 4 mL of PRP will be injected together with 3 +/- 1.5 mL BMAC into the subcortical region of the both ovaries as transvaginal ultra sound guided injection.

After the procedure, during one year follow up, hormone levels of follicle stimulating hormone (FSH), luteinizing hormone (LH),estradiol (E2), progesterone (PG) and anti-mullerian hormone (AMH) would be measured and the follicle numbers would be monitored to provide insight regarding the ovarian function.To investigate the changes in hormone levels, comparisons of the levels detected prior to the intervention, and 3, 6 and 12 months post-intervention, would be performed using Wilcoxon's rank test. Descriptive statistics will be provided for each variable as mean or median number, frequency, percentage, table or graph.

In patients with oocytes retrieved after SEGOVA procedure, standard In Vitro Fertilization protocol would be performed,and fertilization, cleavage and clinical pregnancy rates will be monitored.

ELIGIBILITY:
Inclusion Criteria:

Confirmed informed consent, signature and date

* A woman over 25 years of age
* Primary or secondary amenorrhea for at least 3 months
* Hormone Anti Mullerian Hormone values <_0.42 ng / ML and Follicle stimulating hormone FSH> 20 IU / L, and / or failure of previous attempts of assisted reproductive techniques due to limited ovarian response (less than 3 oocyte cells obtained).
* The proper karyotype 46, XX.
* Presence of at least one ovary

Exclusion Criteria:

* Currently pregnancy or breastfeeding
* Presence of Sexually Transmitted Disease (STD positive)
* There is presence of acute infection (C Reactive Protein>5)
* There is an anamnesis or evidence of existing gynecological malignancy
* The presence of adnexal masses indicating the need for further evaluation.
* It has a contraindication to laparoscopic surgery and / or general anesthesia
* Over the past two weeks, use of the following medicines: Oral or systemic corticosteroids, hormones (estrogen, progestins, oral contraceptives), Danazol, anticoagulants, herbal or botanical supplements with potential hormonal effects.
* Type I diabetes mellitus
* Known significant anemia (hemoglobin <8 g / dL), Severe venous thrombosis and / or pulmonary embolism, Cerebrovascular disease, Presence of heart disease, Premature kidney disease (defined as urea in the blood> 30 mg / dL or serum creatinine> 1.6 mg / dL).

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The eligible patients are women with at least one ovary present.
Enrollment: 100 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Oocyte presence | 12 months
  The numbers of oocytes retrieved after the treatment would be monitored during sonographic follow-ups .
Changes in Hormone Levels of Follicle-stimulating hormone FSH (mIU/mL) | 12 months
  Changes in hormonal levels of FSH toward normal ranges would be monitored during one year follow-up procedure.
Changes in Hormone Levels of Luteinizing Hormone (mIU/mL) | 12
  Changes in hormonal levels of LH toward normal ranges would be monitored during one year follow-up procedure.
Changes in Hormone Levels of Estradiol E2 (pg/mL) | 12
  Changes in hormonal levels of E2 toward normal ranges would be monitored during one year follow-up procedure.
Changes in Hormone Levels of Progesterone PG (ng/mL) | 6
  Changes in hormonal levels of PG toward normal ranges would be monitored during one year follow-up procedure.

SECONDARY OUTCOMES:
Fertilization and implantation rate | 12 months
  Following the Ovarian Rejuvenation Treatment, subjects with oocytes retrieved will undergo IVF protocol, and fertilization and cleavage of embryo would be monitored to evaluate fertility outcomes after SEGOVA procedure.
Number of participants with Positive Clinical Pregnancy | 24 months
  Following completion of trial procedure, patients will be monitored for ongoing clinical pregnancies and conceptions, at the site or via post-treatment correspondence.
Changes in total score of The World Health Organization Quality of Life (WHOQOL) BREF modified scale | 12 months
  Change in quality of life total score for each participant post-procedure would be examined and compared to pre-procedure status. The WHOQOL bref questionnaire would be used as a self-report measure of functional health and well-being. Original WHOQOL bref scale uses 26 questions, while our modified version was abbreviated to 18 questions. The WHOQOL-BREF is scored using a Likert scale, with patients choosing to express how much they agree or disagree with a particular statement from 1 to 5 on a response scale. The value 5 indicates they strongly agree, while 1 is disagree. Total score would be obtained as the sum of 18 questions values from 1 to 5, giving minimum value of total score 18, and a maximum score 90.
Changes in anti-Mullerian hormone (AMH) levels (ng/mL) | 6 months
  Changes in AMH levels would be monitored during one year follow-up procedure and compared to the pre-procedure levels.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandar Ljubic, MD, PhD, Principal Investigator — Medigroup, Belgrade, Serbia
Locations (3):
- Saint James Hospital Malta, Sliema, Malta
- Re-medika Hospital, Skopje, Macedonia, North Macedonia
- Medigroup Health System, Jevremova hospital, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
the individual participant data would be available considering Draft Study Protocol, Statistical analysis Plan, and Informed Consent Forms, and also the data that are published related to this study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Draft study protocol and Statistical Analysis Plan are available entire duration of the study. Informed Consent Forms would be available upon study completion date.
Access Criteria: Access to any additional supporting information about the protocol description or methods used to collect the data will be shared if required by other research organisations. Request would be reviewed by Principal Investigator.
URL: https://segova.com/

REFERENCES:
- [Derived] Tinjic S, Abazovic D, Ljubic D, Vojvodic D, Bozanovic T, Ibrisimovic M, Markovic S, Ljubic A. Influence of Autologous In Vitro Activation of Ovaries by Stem Cells and Growth Factors on Endocrine and Reproductive Function of Patients with Ovarian Insufficiency-A Clinical Trial Study. Int J Fertil Steril. 2021 Jul;15(3):178-188. doi: 10.22074/IJFS.2020.134678. Epub 2021 Jun 22. PMID 34155864